CLINICAL TRIAL: NCT04732689
Title: Intraoperative Hemodynamic Management and Postoperative Outcomes in Liver Transplantation: a Multicenter Prospective Cohort Study
Brief Title: Intraoperative Hemodynamic Management and Postoperative Outcomes in Liver Transplantation
Acronym: ELIPTO-2
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Toronto General Hospital (Other); London Health Sciences Centre (Other); University of Alberta (Other); Queen Elizabeth II Health Sciences Centre (Other); Hopital Paul Brousse (Other); Pitié-Salpêtrière Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20.353
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Liver Failure; Liver Diseases; Surgery; Surgery--Complications; Transplant; Failure, Liver
MeSH Terms: conditions — Liver Failure; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups/Cohorts: The investigators propose to conduct a prospective observational cohort which will include all consecutive adult liver transplant recipients in each center during a one-year period but will exclude same patients who undergo a retransplantation during the same period of observation.

SUMMARY:
The overarching objective of the research program entitled ELIPTO (Enhancing Liver Insufficiency and Postoperative Transplantation Outcomes) (www.elipto.ca) is to improve the perioperative care of liver transplant recipients. One of this program's purposes is to better define the effects of intraoperative hemodynamic management on postoperative outcomes in adult liver transplant recipients. In this study, the incidence of postoperative complications within this population will be defined in Canada and France and the association between intraoperative hemodynamics and postoperative outcomes will be measured.

Liver transplantation improves the survival of patients with end-stage liver disease (ESLD). It is the second most transplanted organ with a continuously increasing annual number of transplantations, an observation partly explained by an endemic ESLD etiology in the United States, the obesity-related non-alcoholic steatohepatitis (NASH) cirrhosis. In recent decades, although sicker patients are prioritized, survival has improved possibly through an overall improvement in the quality of care. However, postoperative complications have concomitantly increased. On average, liver transplant recipients suffer from more than three postoperative complications, mainly infectious, pulmonary, renal or graft-related, two thirds of them being severe. In a low-risk patients cohort, close to 60% of all patients suffered from at least one severe complication up to 6 months after surgery. Such complications increase mortality, readmissions and cost of care. Organs available for transplantation are a scarce resource; up to 10% of grafts are no longer functional after one year. Interventions that improve patients' postoperative and graft outcomes are needed and few perioperative ones are supported by high-quality evidence.

DETAILED DESCRIPTION:
OBJECTIVES:

The main objective of this study is to describe and measure the effects of intraoperative hemodynamic management on postoperative outcomes in liver transplantation in Canada and France.

The specific objectives are:

1. To describe the overall incidence of postoperative complications and graft outcomes in adult liver transplant recipients in Canada and France and across different recipients' characteristics.
2. To measure the effects of fluid balance, within an overall hemodynamic instability and management strategy, on the postoperative outcomes of liver transplant recipients in Canada and France.

The central hypotheses of this study are that an intraoperative hemodynamic management based on a restrictive fluid administration may improve postoperative outcomes in this population.

EXPOSURE VARIABLES:

The exposures of interest will be the intraoperative fluid balance and the intraoperative doses and types of vasopressors used. Fluid balance will be defined as the sum of the volume of administered crystalloids, colloids and blood product transfusions minus drained ascites, intraoperative diuresis and bleeding. Doses of administered vasopressors will be converted into a time-weighted total norepinephrine equivalent dose calculated as the total equipotent units of norepinephrine administered as an infusion divided by the number of hours the infusion was given during the period between entrance in the operating room and end of surgery. Types of vasopressors used will also be collected. Since a restrictive fluid management strategy is associated with a higher use of vasopressors and vice versa, both variables may covary together. However, more difficult surgeries will be associated with higher blood loss, higher volume of administered fluid and higher doses of vasopressors. The combination of these two variables will help estimate the intraoperative hemodynamic management strategy used and delineate the effects of each component.

OTHER DESCRIPTIVE VARIABLES:

Other patients' characteristics and perioperative practices variables will be captured for descriptive purposes. Recipients' demographic characteristics (age, sex), anthropometric variables (body mass index (BMI)), the presence of any previous abdominal surgery, presence of hepatic encephalopathy, need for preoperative organ support or any preoperative hospital admission will be collected as well. Data on the perioperative use of invasive cardiac output monitoring (thermodilution catheter, transoesophageal echocardiography, etc.), as well as coagulation management (use of thromboelastometry, tranexamic acid, transfusion thresholds, etc.) will be collected. Other donor and graft variables, such as donor sex, donor's BMI, the type of vascular and biliary anastomoses, the use of extended-criteria donor graft, the use of ex vivo perfusion, ischemia time, the practice of donation after circulatory death (donor characteristics, heparin usage, etc.) and the perioperative use of liver biopsies will also be collected.

DESCRIPTIVE AND STATISTICAL ANALYSIS:

Missing data The investigators will train all sites regarding quality of data collection and will emphasize the importance of complete data collection. In case a complete case analysis would exclude more than 5% of the observations, the investigators will use multiple imputations by chained equations using 5 to 20 imputated datasets assuming MAR (missingness at random) on the covariables and the outcomes.

Descriptive analyses and complications incidences across centers The investigators will first describe the cumulative incidences of different complications or categories of complications as previously defined. Their main descriptive analysis will be to report these incidences overall as well as across denominated centers. Then, they will estimate multivariable determination models for each complication category by fitting generalized mixed effect models using a logit link adjusted for age, sex, disease severity (MELD), transplantation indication, requirement for preoperative organ support and donor characteristics with an estimated random-effect for clustering within centres. The investigators will then compute intra-class correlation (ICC) coefficients to better define the variability of complications across centres (heterogeneity). However, they will fit a Cox regression with a shared frailty factor for biliary complications. Finally, they will fit a generalized mixed effect model using a log link and quasi-Poisson distribution for the total number of complications up to 30 days per patient with an estimated random effect for clustering within centres. Their secondary exploratory analyses will be to report the cumulative incidence of each complication according to age categories (< 50, 50-60, >60), sex, nature and severity of liver disease (chronic liver disease (CLF), acute liver failure (ALF), retransplantation and MELD categories among CLD patients (< 20, 20-30, >30). They will report such incidences per subgroups with 95% confidence intervals. They will also report survival up to 6 months over and across centres by fitting a Cox regression with a frailty factor.

Association between hemodynamic management and postoperative complications The investigators' primary analysis will be the association between fluid volume and primary graft dysfunction by 7 days after transplantation using a multivariable generalized mixed-effect model using a logistic link and random intercepts, adjusted for the time-weighted dose of vasopressors and the aforementioned confounders, and estimated using residualized penalized quasi-likelihood. They will consider any patient needing a retransplantation within 7 days after the index transplantation as having a primary graft dysfunction. Statistical interaction will be explored between fluid balance and the vasopressors dose variable.

The investigators' other secondary analyses will be the association between fluid volume and other outcomes, including AKI and the total number of complications up to 30 days, using similar adjusted survival models (with frailty factors) or generalized mixed effect models (with random intercepts). Among them, the investigators will analyze the association between fluid volume and time to biliary non-anastomotic strictures using a multivariable Fine and Gray model, adjusted for the same confounders, with retransplantation and death (not caused by the biliary non-anastomotic strictures) considered as competing risks. They will address intra-cluster correlation using a frailty factor. Risk proportionality over time will be explored using the Harrel and Lee test and a visual inspection of the Schoenfeld residuals.

Subgroup analysis The investigators will conduct a subgroup analysis comparing the effect of their exposures on the primary outcome in the subgroup of patients transplanted for end-stage liver disease and those transplanted for causes other than end-stage liver disease. The investigators will thus estimate the same model but with an interaction term between the fluid volume and a dummy variable for end-stage liver disease. They will report stratified results with 95% CI and the interaction test p value.

Sensitivity analyses For the primary outcome, the main secondary outcome and the total number of complications at 30 days, the investigators will first conduct a sensitivity analysis using a generalized propensity score for fluid volume (based on probability density) that will include all confounders and the vasopressor exposure and estimate a marginal effect of fluid balance using an inverse probability of treatment weighting with stabilized weights. The investigators will evaluate the confounding effect of hypotension by removing it from the models as well as by a sensitivity analysis restricted in the subgroup of patients without significant residual hypotension. Finally, they will conduct all analyses by adding data from the French centre to explore the variation in the estimates created by adding a non-Canadian centre.

Economic analysis The investigators will conduct an economic analysis to evaluate hospital costs associated with the observed incidences of postoperative complications. They will also analyze costs associated with their fluid balance exposure effect. Costs will be those associated with the actual procedures, as determined by every hospital using its account systems, and include both fixed and variable components previously identified as major cost drivers (mechanical ventilation days, LOS, reoperation and ICU readmission).

ELIGIBILITY:
Inclusion Criteria:

All consecutive adult liver transplant recipients in each center during a one-year period or more (anywhere in between June 1, 2021 and November 30, 2022).

Exclusion Criteria:

Same patients who undergo a retransplantation during the same period of observation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The investigators will include all recipients of a liver transplant across six Canadian centres, as well as in one French Centre.
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Occurence of primary graft dysfunction | At 7 days after transplantation
  This outcome was chosen because preliminary data from the CHUM suggested that a higher fluid balance was associated with primary graft non-function (retransplantation or death). Since graft perfusion is correlated with cardiac output, intraoperative hemodynamic management may have an effect on graft perfusion and postoperative graft function. Also, this is a well-defined, quantitative definition, that is associated with overall graft and patient survival. Since graft loss of 10% at 1 year is a concern among the transplant community, finding causes and solutions to improve graft function is paramount.

SECONDARY OUTCOMES:
Occurrence of biliary complications | Up to 6 months after transplantation
  Biliary complications have major impacts on patients' quality of life, graft survival and mortality. While biliary ducts are sensible to ischemic injury, the incidence of non-anastomotic strictures have been overlooked in previous perioperative studies. Biliary complications will be classified as any stricture (anastomotic or non-anastomotic) based on medical imaging results and/or surgical, endoscopic and radiological procedures.
Occurence of biliary anastomotic strictures | Up to 6 months after transplantation
  Biliary complications will be classified as any stricture (anastomotic or non-anastomotic) based on medical imaging results and/or surgical, endoscopic and radiological procedures.
Liver transplant-related reoperations | Up to 30 days after transplantation
  Patient having to undergo any liver transplant-related reoperations up to 30 days after transplantation.
Retransplantation | Up to 6 months after transplantation
  Retransplantation is defined as the patient having to undergo a new transplantation following the index transplantation.
Occurence of acute kidney injury | 48 hours, 7 days and 30 days after transplantation
  The grade of AKI was classified according to the KDIGO-AKI criteria using the highest reported creatinine or the need for new renal replacement therapy after surgery, including any mode of renal replacement therapy.
Occurence of infectious complications | Up to 30 days after transplantation
  Infectious complications by any antibiotic prescription lasting more than 72 hours
Occurrence of pulmonary complications | Up to 30 days after transplantation
  Pulmonary complications will be classified using standardized definitions for atelectasis and ARDS.
The need for a new postoperative ICU admission | Up to 30 days after transplantation
  The dates for all ICU admissions and dates of ICU discharge were recorded. If the patient was readmitted to ICU following his initial admission to ICU, the dates for admissions and discharges were recorded.
30-day mechanical ventilation free-days | Up to 30 days after transplantation
  The total number of days the patient was on invasive mechanical support was recorded. If mechanical ventilation was weaned and started again, the days when the patients were under mechanical ventilation were indicated. Non-invasive ventilation or high-flow nasal cannula (HFNC) were not included.
30-day organ dysfunction free days | Up to 30 days after transplantation
  The total number of days the patient was: on invasive mechanical ventilator, under vasopressor therapy for more than 2 hours up to 30 days after surgery and spent under renal replacement therapy was recorded.
Hospital length of stay | 30 days after transplantation
  The number of days of hospital length of stay was calculated using the difference between the local date of discharge from the hospital and the date of hospital admission (day of surgery). If the patient died during surgery or prior to hospital discharge, the patient's date of death was recorded as the date of discharge.
Occurence of acute rejection episode | 30 days after transplantation
  An acute rejection episode defined as the grafted liver is attacked by the immune system.
Survival up to 6 months | 6 months after transplantation
  Survival was calculated from the date of participant initial transplant to the date of participant death due to any cause, within 6 months after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: François-Martin Carrier, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided